CLINICAL TRIAL: NCT06069258
Title: Movement Behaviours Among Bahraini Type 2 Diabetic Adults: a Cross-sectional Study
Brief Title: Movement Behaviours Among Bahraini Diabetics
Status: Recruiting | Type: Observational
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: Ministry of Health, Bahrain (Other Government); Arabian Gulf University, Bahrain (Other); Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Other Study IDs: 284/23-Oct-222
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Physical activity; Behaviour; mHealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bahraini adults with type 2 diabetes: Male and female Bahraini adults aged 20-75 years with controlled type 2 diabetes (i.e. HbA1c <9 on medication).

SUMMARY:
This observational study aims to measure movement behaviours and explore factors influencing these among Bahraini patients with type 2 diabetes.

The main objectives are:

(i) Measure free-living physical activity and sedentary behaviour with an accelerometer device (ii) Examine associations between movement behaviours and anthropometric and diabetes-related biochemical/clinical parameters (iii) Examine associations between movement behaviours and psychological and environmental determinants that influence movement behaviours (iv) Assess the feasibility and acceptability of the physical activity assessment tools as part of routine clinical practice with clinicians and diabetic patients

Participants will be invited to wear an accelerometer device for seven days.

DETAILED DESCRIPTION:
In Bahrain, the number of people diagnosed with diabetes has risen from 9% at the start of the new millennium to 15% in 2022, and like any other country, it places a significant burden on the country's health system. People with type 2 diabetes mellitus (T2DM) are more sedentary, do less physical activity (PA), have lower cardiovascular fitness levels and are at higher risk for comorbid conditions that may affect mobility (e.g., sarcopenia and diabetic foot ulcers) compared to people without diabetes. Regular aerobic physical activity benefits in this clinical population include reduced HbA1C, triglycerides, blood pressure, body fat, and insulin resistance. Understanding the PA and sedentary behaviour patterns of Bahraini adults with T2DM is an essential first step towards our long-term goal of planning and developing a physical activity intervention.

A combination of self-efficacy and outcome expectations influence behaviour change, and it is important to understand the relationship between these in any specific T2DM population to identify appropriate interventions. Improving uptake and adherence to PA by people with T2DM also requires an understanding of any enablers and barriers.

This study aims to measure movement behaviours among Bahraini adult patients with T2DM using an accelerometer device and to examine associations with anthropometric and biochemical/clinical parameters, psychological and environmental determinants that influence these behaviours, and to assess the feasibility and acceptability of the PA assessment tools as part of standard clinical practice with clinicians and people with diabetes.

The study design will be observational and conducted at four specialist government diabetic clinics drawn from across the governorates of Bahrain. We aim to recruit 320 Bahraini adults 45-64 years old with controlled T2DM.

Participants will attend two visits seven days apart:

Visit 1: Anthropometric measurements will be conducted. information on sociodemographic characteristics will be collected. Information on select clinical parameters will be collected from the medical record of each patient's last visit to the health centre for routine follow-up within the last four months; otherwise, these measurements will be ordered. Participants will complete questionnaires to investigate behavioural and environmental determinants of physical activity. Participants will be fitted with an accelerometer device (activPALTM) and advised to wear it for the next seven days, after which they should return for visit 2. Finally, each participant will receive an activity diary to complete each day.

Visit 2: Participants will return the accelerometer and activity diary. They will also complete the same questionnaires of behavioural and environmental determinants which were administered in visit 1. Finally, participants will complete a utility questionnaire about the accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Men and women are eligible.
* Age: Individuals aged 20-75 years old are eligible.
* Ethnicity: Bahraini adults of all ethnic groups are eligible for the study.
* Type 2 diabetes and glycaemic control: Individuals with controlled type 2 diabetes (i.e. HbA1c <9 on medication) based on the medical record of each patient's last visit to the health centre for routine follow-up will be eligible if within the last four months. Otherwise, these measurements will be ordered at the first visit to confirm eligibility.
* Blood pressure: Individuals whose blood pressure is under moderate control will be eligible - specifically, treated or untreated resting systolic/diastolic pressure < 160/100 mmHg.
* Lipid control: Individuals with fasting triglyceride concentration < 600 mg are eligible.

Exclusion Criteria:

* HbA1c >9%
* Type 1 diabetes
* Taking insulin
* Pregnancy
* Non-ambulant or severely incapacitated with any medical condition(s) reducing ability to stand or mobilize.
* Currently participating in a study to reduce sedentary behaviour or increase physical activity
* Language. Inability to read and understand Arabic or English language.
* Inability to give informed consent.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bahraini adults of all ethnicities with controlled diabetes.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Movement behaviour | 1 week (duration of the study)
  Movement behaviour will be assessed using a thigh-worn accelerometer (activPAL, PAL Technologies, Scotland, U.K. www.palt.com). It has no screen to indicate the amount of physical activity being done, so does not act as a motivational device. The activPAL will be used to collect data 24 hours/day over seven consecutive days.

SECONDARY OUTCOMES:
Activity diary | 1 week (duration of the study)
  Participants will also be asked to keep an activity diary to record when they got up from and went to bed, took part in any activities, or when and why they removed the device.
Sociodemographic characteristics | Day 1/baseline
  Baseline data for age, gender, educational level, marital status, occupation, and type of living accommodation (or living arrangements) will be obtained by a self-administered questionnaire to describe the sample recruited at the start of the study.
Anthropometric parameters | Day 1/baseline
  Baseline data for body weight status and fat distribution will be established using the standard measurements of body mass index (BMI), waist circumference, and waist-to-hip ratio. Body Mass Index (BMI) will be calculated as weight divided by the square of the height (kg/m2). Standard categories of body weight status will be applied (underweight: <18.50 kg/m2; normal weight: 18.50-24.99 kg/m2; overweight: 25.00-29.99 kg/m2; obese: ≥30.00 kg/m2). Waist circumference >102 cm for men and >88 cm for women will be classified as having abdominal obesity. Waist-to-hip ratios of ≥0.9 and ≥0.9 for men and ≥0.8 and ≥0.85 for women will be classified as overweight and obese, respectively.
Clinical parameters | Day 1/baseline
  Blood pressure, diabetes duration, smoking status, low-density lipoprotein (LDL), glycated haemoglobin (HbA1c), estimated glomerular filtration rate (e-GFR), and medication will be collected from the medical record of each patient's last visit to the health centre for routine follow-up if within the last four months. Otherwise, these parameters will be ordered at the first visit.
Exercise Self-Efficacy | Day 1/baseline and end of study (day 7)
  Self-efficacy will be investigated using the Exercise Self-Efficacy Scale, which has been validated and is available in English and Arabic. The questionnaire consists of nine items, each of which is scored between zero (not confident) to ten (very confident). The total score is calculated by summing the responses to each question. A higher score indicates higher self-efficacy for exercise. Participants will complete this questionnaire at the start/baseline and end of the study.
Motivation to Exercise | Day 1/baseline and end of study (day 7)
  Motivation to exercise will be investigated using the Behavioral Regulation in Exercise Questionnaire (BREQ-3). This multidimensional instrument consists of 24 items with a five-point Likert Scale and a separate score for each of the subscales (amotivation, external regulation, introjected regulation, identified regulation, integrated regulation and intrinsic motivation). This instrument is valid, and reliable and is available in English and Arabic (13). Participants will complete this questionnaire at the start/baseline and end of the study.
Factors affecting movement behaviour | Day 1/baseline and end of study (day 7)
  Factors influencing movement behaviour will be investigated using our modified version of the Capability, opportunity and Motivation (COM-B) questionnaire (14), called the Physical Activity Behaviour Self Evaluation Questionnaire, which consists of 22 items. Participants will complete this questionnaire at the start/baseline and end of the study.
Wearability of the ActivPAL device | Day 7
  A utility questionnaire will be used to facilitate feedback from participants about the ActivPAL activity monitor. The questions include a 10-point visual analogue scale from (0) 'very difficult/uncomfortable' through to (10) 'very easy/comfortable' to assess the ease of fitting and comfort of wearing the ActivPAL device. Participants will also be asked to comment on any difficulties wearing the monitors or any strategies they adopted to make it easier to wear them.
Adverse events | Duration of the study and up to two weeks afterwards
  A standard adverse events form will be used to record any significant issues for participants due to the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrahim Rajab, PhD, Principal Investigator — Royal College of Surgeons in Ireland - Medical University Bahrain
Locations (4):
- Bahrain (4):
  - Isa Town Health Centre, Building 10, Road 43, Manama
  - Ahmed Ali Kanoo Health Centre, Building 2009, Road 2641, Manama
  - Halat Bu Maher Health Centre, Building 2858, Road 1653, Muharraq
  - Shaikh Jaber AlSabah Health Centre, Building 6347, Road Nakheel Street, Northern Governorate

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available all de-identified IPD that underlies results in the publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted 6 months after article publication, and the data will be accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in diabetes and physical activity. To gain access, requestors will need to sign a data access agreement.